CLINICAL TRIAL: NCT04486313
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled, Trial to Evaluate Efficacy and Safety of Nitazoxanide in the Treatment of Mild or Moderate COVID-19
Brief Title: Trial to Evaluate Efficacy and Safety of Nitazoxanide in the Treatment of Mild or Moderate COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM08-3008
Record Dates: First submitted 2020-07-23; First posted 2020-07-24 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Active Comparator): Two nitazoxanide 300 mg tablets orally twice daily for 5 days
  Interventions: Drug: Nitazoxanide; Dietary Supplement: Vitamin Super B-Complex
- Placebo (Placebo Comparator): Two placebo tablets orally twice daily for 5 days
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin Super B-Complex

INTERVENTIONS:
Drug: Nitazoxanide — Two nitazoxanide 300 mg tablets administered orally twice daily with food for 5 days
  Other Names: NTZ (nitazoxanide); NT-300
  Arms: Nitazoxanide
Drug: Placebo — Two placebo tablets administered orally twice daily with food for 5 days
  Arms: Placebo
Dietary Supplement: Vitamin Super B-Complex — Vitamin Super B-Complex administered orally twice daily to maintain the blind

SUMMARY:
Trial to Evaluate Efficacy and Safety of Nitazoxanide in the Treatment of Mild or Moderate COVID-19

DETAILED DESCRIPTION:
Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Efficacy and Safety of Nitazoxanide in the Treatment of Mild or Moderate COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 12 years of age
* Presence of clinical signs and/or symptoms consistent with worsening or stable mild or moderate COVID-19 (one of the following is required):

  1. Presence of at least two respiratory symptom domains (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO OR
  2. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO with pulse rate ≥90 OR
  3. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO with respiratory rate ≥16

AND patient reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day, as confirmed by responses to questions in the Screening FLU-PRO.

* Onset of symptoms no more than 72 hours before enrollment in the trial. Onset of symptoms is defined as the earlier of the first time at which the subject experienced subjective fever or any respiratory symptom (head, throat, nose, chest, or cough symptoms).
* Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the subject diary and all protocol procedures.

Exclusion Criteria:

* Persons with any clinical sign or symptoms suggestive of severe systemic illness with COVID-19, including the following:

  1. shortness of breath at rest,
  2. resting pulse ≥125 beats per minute,
  3. resting respiratory rate ≥30 breaths per minute, or
  4. SpO2 ≤ 93% on room air at sea level.
* Subjects who experienced a previous episode of acute upper respiratory tract infection, otitis, bronchitis or sinusitis or received antibiotics for these conditions within two weeks prior to and including study day 1.
* Severely immunodeficient persons including:

  1. Subjects with immunologic disorders or receiving immunosuppressive therapy (e.g., for organ or bone marrow transplants, immunomodulatory therapies for certain autoimmune diseases)
  2. Subjects with untreated human immunodeficiency virus (HIV) infection or treated human immunodeficiency virus (HIV) infection with a CD4 count below 350 cells/mm3 in the last six months
  3. Subjects actively undergoing systemic chemotherapy or radiotherapy treatment for malignancy
  4. Subjects using steroids as maintenance therapy for chronic conditions
* Subjects with active respiratory allergies or subjects expected to require anti- allergy medications during the study period for respiratory allergies.
* Females of childbearing potential who are either pregnant or sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an intrauterine device (IUD), or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year - or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral oophorectomy.
* Subjects with a history of COVID-19 or known to have developed anti-SARS- CoV-2 antibodies.
* Subjects residing in the same household with another subject participating in the study.
* Treatment with any investigational drug or vaccine therapy within 30 days prior to screening and willing to avoid them during the course of the study.
* Receipt of any dose of nitazoxanide within seven days prior to screening.
* Known sensitivity to nitazoxanide or any of the excipients comprising the study medication.
* Subjects unable to swallow oral tablets or capsules.
* Subjects with known severe heart, lung, neurological or other systemic disease that the Investigator believes could preclude safe participation.
* Subjects likely or expected to require hospitalization unrelated to COVID-19 during the study period.
* Subjects taking medications considered to be major CYP2C8 substrates.
* Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol including completion of the subject diary.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 935 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Invesclinic US LLC, Fort Lauderdale, Florida
  - RH Medical Urgent Care, The Bronx, New York

REFERENCES:
- [Derived] Rossignol JF, Bardin MC, Fulgencio J, Mogelnicki D, Brechot C. A randomized double-blind placebo-controlled clinical trial of nitazoxanide for treatment of mild or moderate COVID-19. EClinicalMedicine. 2022 Feb 28;45:101310. doi: 10.1016/j.eclinm.2022.101310. eCollection 2022 Mar. PMID 35237748

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitazoxanide | Placebo
Started | 472 | 463
Completed | 453 | 446
Not Completed | 19 | 17
Not completed — Lost to Follow-up | 7 | 9
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Death | 2 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide | Placebo | Total
Number analyzed (Participants) | 472 | 463 | 935
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (14.83) | 40.7 (14.68) | 40.5 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 284 | 566
  Male | 190 | 179 | 369
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 117 | 112 | 229
  Not Hispanic or Latino | 349 | 343 | 692
  Unknown or Not Reported | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 6 | 5 | 11
  Black or African American | 41 | 43 | 84
  White | 404 | 388 | 792
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 14 | 19 | 33
Height [Mean (Standard Deviation); unit: centimeters] | 169.1 (10.84) | 168.4 (9.96) | 168.7 (10.41)
Weight [Mean (Standard Deviation); unit: kilograms] | 88.0 (24.44) | 88.5 (23.36) | 88.3 (23.90)
BMI [Mean (Standard Deviation); unit: kilograms per meters squared] | 30.7 (7.72) | 31.1 (7.51) | 30.9 (7.62)
Time from Onset of Symptoms to Randomization [Mean (Standard Deviation); unit: hours] | 41.5 (15.73) | 41.9 (16.71) | 41.7 (16.21)
Tobacco Use [Count of Participants; unit: Participants]
  Current Tobacco User | 115 | 106 | 221
  Past Tobacco User | 62 | 69 | 131
  Never Used Tobacco | 295 | 288 | 583
Severity of Disease [Count of Participants; unit: Participants] — Baseline illness severity was defined as follows:
  Mild illness: resting pulse <90 beats per minute and resting respiratory rate <20 breaths per minute.
  Moderate illness: resting pulse ≥90 beats per minute or resting respiratory rate ≥20 breaths per minute.
  Participants
    Mild Illness | 301 | 305 | 606
    Moderate Illness | 170 | 158 | 328
    Unknown | 1 | 0 | 1
Risk of Severe Illness [Count of Participants; unit: Participants] — Risk was defined as follows according to data published by CDC:
  At Increased Risk: Subjects with COPD, Type 2 diabetes mellitus, obesity (BMI ≥30), chronic kidney disease, sickle cell disease, serious heart conditions, asthma (moderate or severe), cerebrovascular disease, cystic fibrosis, hypertension or high blood pressure, immunocompromised state, neurologic conditions, liver disease, pulmonary fibrosis, past or present history of smoking, thalassemia, or type 1 diabetes mellitus. Subjects who are ≥65 years of age.
  Not at Increased Risk: Subjects with none of the above conditions
  Participants
    At Increased Risk of Severe Illness | 330 | 338 | 668
    Not At Increased Risk of Severe Illness | 142 | 125 | 267

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Clinical Recovery
Description: Time to Sustained Clinical Recovery is the time in days from the first dose of study medication to the first time at which the subject reports a decrease in total FLU-PRO score from the previous diary with assessment that symptoms are at least "somewhat better than yesterday", no oral temperature ≥100.4 F in the prior 24 hours, and no future increase in any of the FLU-PRO domains except within validated background levels.
Time Frame: Up to 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for SARS-CoV-2 by RT-PCR at Baseline.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 184 | 194
days | 13.3 [6.26 to 21] | 12.4 [7.18 to 21]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.8786, Gehan-Wilcoxon Test; Stratified by Baseline COVID-19 severity (mild/moderate), time from onset of symptoms to randomization (<36 hours/≥36 hours), risk of severe illness

2. Secondary Outcome: Proportion of Subjects Progressing to Severe COVID-19
Description: Analysis of proportions of subjects with progression to severe COVID-19 illness defined as subject-reported shortness of breath at rest and blood oxygen saturation ≤93% on room air
Time Frame: Up to 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for SARS-CoV-2 by RT-PCR
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 184 | 195
proportion of subjects | 0.005 | 0.036
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.0740, Cochran-Mantel-Haenszel — Stratified by Baseline COVID-19 severity (mild/moderate), time from onset of symptoms to randomization (<36 hours/≥36 hours), risk of severe illness

3. Other Pre Specified Outcome: Proportion of Subjects Positive for SARS-CoV-2 by Aptima® SARS-CoV-2 Assay at Each of Days 4 and 10
Time Frame: Day 4 and Day 10
Population: The ITTI (primary efficacy) population consisted of all subjects positive for SARS-CoV-2 by RT-PCR
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 184 | 195
proportion of subjects
  Day 4 | 0.908 | 0.862
  Day 10 | 0.707 | 0.662
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Comparison of proportion positive for SARS-CoV-2 at Day 4; Test type: Superiority; p = 0.4479, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Nitazoxanide vs Placebo; Comparison of proportion positive for SARS-CoV-2 at Day 10; Test type: Superiority; p = 0.2814, Cochran-Mantel-Haenszel

4. Other Pre Specified Outcome: Change From Baseline in Quantitative SARS-CoV-2 RNA Measured by RT-PCR at Each of Days 4 and 10
Time Frame: Day 4 and Day 10
Population: The ITTI (primary efficacy) population consisted of all subjects positive for SARS-CoV-2 by RT-PCR
Measure: Mean (Standard Error); unit: log10 RNA copies/milliliter
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 184 | 195
log10 RNA copies/milliliter
  Day 4 | -0.70 (0.118) | -1.02 (0.126)
  Day 10 | -2.49 (0.119) | -2.61 (0.120)
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Comparison of change from Baseline to Day 4; Test type: Superiority; p = 0.0665, t-test, 2 sided
Statistical Analysis 2: Comparison: Nitazoxanide vs Placebo; Comparison of change from Baseline to Day 10; Test type: Superiority; p = 0.4974, t-test, 2 sided

5. Other Pre Specified Outcome: Proportion of Subjects Requiring Hospitalization
Description: Analysis of proportions of subjects requiring hospitalization for any reason during the study period
Time Frame: 28 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for SARS-CoV-2 by RT-PCR
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 184 | 195
proportion of subjects | 0.005 | 0.026
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.1771, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

6. Other Pre Specified Outcome: All-Cause Mortality
Description: Analysis of proportions experiencing mortality from any cause during the study period
Time Frame: 28 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for SARS-CoV-2 by RT-PCR
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 184 | 195
proportion of subjects | 0.005 | 0.000
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.2399, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

7. Post Hoc Outcome: Time to Sustained Recovery for Subjects With Mild Illness
Description: as for outcome 1
Time Frame: 21 days
Population: The ITTI (primary efficacy) population consisted of all subjects positive for SARS-CoV-2 by RT-PCR. Mild illness is defined as subjects with pulse <90 beats per minute and respiratory rate <20 breaths per minute at Baseline.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 116 | 130
days | 10.3 [6.2 to 21] | 13.4 [7.4 to 21]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.09, Gehan-Wilcoxon Test; [statistical method as in outcome 1, analysis 1]

8. Post Hoc Outcome: Time to Return to Usual Health for Subjects With Mild Illness
Description: Subjects completed a diary daily in the evening. The time from first dose to ability to return to usual health is the time in days from the first dose of study medication to the first time when the subject answered "Have you returned to your usual health?" with "yes" for two consecutive daily diary periods.
Time Frame: 21 days
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 116 | 130
days | 13.2 [9.2 to 21] | 18.4 [11.4 to 21]
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.0077, Gehan-Wilcoxon Test; [statistical method as in outcome 1, analysis 1]

9. Post Hoc Outcome: Progression to Severe COVID-19 for Subjects At Least Possibly At Increased Risk Per CDC Guidelines
Description: Analysis of proportions of subjects with progression to severe COVID-19 illness defined as subject-reported shortness of breath at rest and blood oxygen saturation ≤93% on room air for the subgroup of subjects considered possibly at high risk per CDC guidelines
Time Frame: 28 days
Population: Subjects positive for SARS-CoV-2 by RT-PCR with one of the following risk factors: COPD, Type 2 diabetes mellitus, obesity (BMI≥30), chronic kidney disease, sickle cell disease, serious heart conditions, ≥65 years of age, asthma (moderate or severe), cerebrovascular disease, cystic fibrosis, hypertension or high blood pressure, immunocompromised state, neurologic conditions, liver disease, pulmonary fibrosis, past or present history of smoking, thalassemia, Type 1 diabetes mellitus
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 112 | 126
proportion of subjects | 0.009 | 0.056
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

10. Post Hoc Outcome: Progression to Severe COVID-19 for Subjects At Increased Risk Per CDC Guidelines
Description: Analysis of proportions of subjects with progression to severe COVID-19 illness defined as subject-reported shortness of breath at rest and blood oxygen saturation ≤93% on room air for the subgroup of subjects considered high risk per CDC guidelines
Time Frame: 28 days
Population: Subjects positive for SARS-CoV-2 by RT-PCR with one of the following risk factors: COPD, Type 2 diabetes mellitus, obesity (BMI≥30), chronic kidney disease, sickle cell disease, serious heart conditions, ≥65 years of age.
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 104 | 121
proportion of subjects | 0.009 | 0.057
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.05, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

11. Post Hoc Outcome: Progression to Severe COVID-19 in Subjects at High Risk by FDA Guidelines
Description: Analysis of proportions of subjects with progression to severe COVID-19 illness defined as subject-reported shortness of breath at rest and blood oxygen saturation ≤93% on room air for the subgroup of subjects considered at high risk per FDA guidelines
Time Frame: 28 days
Population: Subjects positive for SARS-CoV-2 with at least one of the following risk factors: ≥ 65 years of age, BMI ≥35 kg/m2, chronic kidney disease, diabetes, immunosuppressive disease, current receipt of immunosuppressive treatment, or ≥55 years of age with at least one of cardiovascular disease, hypertension, or chronic obstructive pulmonary disease or another chronic respiratory disease.
Measure: Number; unit: proportion of subjects
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 60 | 69
proportion of subjects | 0.016 | 0.086
Statistical Analysis 1: Comparison: Nitazoxanide vs Placebo; Test type: Superiority; p = 0.08, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Nitazoxanide | Placebo
All-Cause Mortality (participants affected / at risk) | 2/472 | 0/463
Serious Adverse Events (participants affected / at risk) | 2/472 | 7/463
Other Adverse Events (participants affected / at risk) | 16/472 | 10/463
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=472) | Placebo (N=463)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=472) | Placebo (N=463)
Diarrhoea (Gastrointestinal disorders) | 16 (472) | 10 (463)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT04486313/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT04486313/SAP_001.pdf